CLINICAL TRIAL: NCT03079778
Title: Transarterial Chemoembolization (TACE) With or Without Stereotactic Body Radiotherapy (SBRT) in Hepatocellular Carinoma
Acronym: TACERT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Opened up a separate Clinicaltrials.gov trial form, study ID TACE
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106681
Record Dates: First submitted 2016-03-11; First posted 2017-03-14 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: randomized to radiation (RT) or TACE plus RT (TACERT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE alone (Active Comparator): Transarterial chemoembolization (TACE)
  Interventions: Procedure: transarterial chemoembolization
- TACE plus RT (Experimental): Combination of transarterial chemoembolization and radiation (TACERT)
  Interventions: Procedure: transarterial chemoembolization; Radiation: TACE plus RT

INTERVENTIONS:
Procedure: transarterial chemoembolization — Transcatheter arterial chemoembolization (also called transarterial chemoembolization or TACE) is a minimally invasive procedure performed in interventional radiology to restrict a tumor's blood supply
Radiation: TACE plus RT — radiobiologically guided radiation
  Other Names: radiobiological guided radiation
  Arms: TACE plus RT

SUMMARY:
Hypothesis: Patients with hepatocellular carcinoma (HCC) have few options if they fail or are unable to undertake surgery, transarterial chemoembolization (TACE) and/or chemotherapy. Radiation (RT) in a range of doses has been combined with TACE in several case cohort studies demonstrating safety and a dramatic improvement in survival. Clearly these trials are subject to bias due to non-randomized selection, possible lack of generalizability to Canadian patients, and heterogeneous patient populations.

Objective: Therefore, there is a high priority need to investigate the addition of RT to TACE in a randomized fashion to determine if we can improve survival in this rapidly growing poor prognosis patient population that have no other options.

Methodology: TACE eligible patients with HCC will be randomized to TACE alone or TACE plus radiation (TACERT). They cannot be eligible for standard treatments such as transplant and resection. Primary endpoint will be time-to-intrahepatic-progression. Secondary endpoints will be response rate (Modified RECIST criteria), overall survival, local failure, extrahepatic failure, toxicity, quality of life and economic feasibility.

DETAILED DESCRIPTION:
DETAILED OUTLINE OF RESEARCH PROPOSAL

Current State of Knowledge Primary liver cancer, hepatocellular carcinoma (HCC), is a major health problem worldwide. It is the 5th most common cancer and the 3rd most common cause of cancer death in the world. Eighty-five percent of cases occur in developing countries, while in the United States and Canada, it is the fastest growing cancer.

General Treatment Overview: HCC tends to remain within the liver and, therefore, cure with preserved liver function is possible. Surgical resection results in 5-year survival rates of 60%-70%. Liver transplantation can cure both the cancer and underlying liver disease. Four-year survival for HCC within the Milan criteria (single HCC <5 cm or ≤3 HCC <3 cm) is 70%-85% after transplantation. Unfortunately, most patients are not resectable. Transarterial chemoembolization (TACE) has become the mainstay of treatment for unresectable HCC. What makes TACE relatively safe is the liver-unique vascular supply from the portal vein, whereas HCC is supplied almost entirely by branches of the hepatic artery. In a randomized controlled trial for unresectable HCC not suitable for a curative intent, transarterial chemoembolisation or TACE were compared to conservative treatment. TACE induced objective responses (complete and partial response) that were sustained for at least 6 months in 35% of cases. Survival probabilities at 1 year and 2 years were 82% and 63% for TACE, significantly better than 63% and 27% obtained with conservative treatment. Overall survival at 1 and 2 years was also significantly better for the chemoembolization group 57% and 31% vs. 32% and 11%. However, many patients have large tumours and response rates decline rapidly with increasing size. TACE alone results in 2 year overall survivals of 42%, 0 and 0 for lesions 5-7cm, 8-10cm, and >10cm, respectively. Therefore, additional locally ablative treatments are being sought. In the same report, TACE plus radiation results in 2 year overall survivals of 63%, 50% and 17% for lesions 5-7cm, 8-10cm, and >10cm, respectively.

External beam radiotherapy has long been considered to have a very limited role in the treatment of liver tumors. This is due to the fact that the minimum dose required for local ablation exceeded the dose that would result in liver toxicity. The technical development of stereotactic body radiation therapy (SBRT), alone or in combination with TACE, renewed interest in radiation for HCC. This work was done mainly by two groups, in Michigan and Stockholm, who demonstrated that the delivery of high doses of radiation to limited volumes of the liver had promising results in terms of local control and survival with acceptable toxicity. Dr. Lock and his team are one of the first centres to initiate this type of work and currently have one of the largest databases outside of asia. In addition, he leads one of only two groups in Canada able to dose escalate based on radiobiological parameters thereby providing the highest possible doses within known toxicity constraints. For SBRT, advanced techniques are used to very accurately deliver a high total dose to the target in a small number of daily fractions while avoiding dose delivery to surrounding healthy structures. SBRT is offered as an ablative radical local treatment. In total, eleven primary series reported on tumor response and survival of around 300 patients who have been treated with stereotactic body radiation therapy as primary therapy for HCC. The reported percentage of objective responses defined as complete and partial was ≥64% in 7 of 8 series. Median survival between 11.7 and 32 months has been observed. Toxicity, based on multiple case series trials, indicate that the treatment is considered safe. The most common CTC grade 3-4 toxicity was elevation of liver enzymes.

For unresectable cases, both TACE and SBRT have been used safely and with good efficacy as separate treatments. Particularly for larger lesions that are more commonly seen in London, the outcome remains suboptimal compared to surgery. Combined treatment case series have shown dramatic results, but there has not been any randomized trial to compare the value of combining the two modalities. Therefore a clinical study comparing SBRT and SBRT+TACE will be significant as it addresses a common problem in one of the two most deadly cancers.

Combined Modality Treatment RT in a range of doses has been combined with TACE in several case cohort studies. One example is a phase 1 dose escalation study that demonstrated that 62 Gy and 52 Gy were safe doses for HCC <10 cm and >10 cm, respectively, in conjunction with TACE. Koo et al prospectively studied 42 patients who received TACE followed by RT. Survival in this cohort was improved compared with a historical control group of 29 patients who received TACE alone (median survival 11.7 vs. 4.7 months). Four studies specifically compared cohorts of patients that received TACE alone versus TACE+SBRT. All demonstrated significant improvement in response rates and overall survival. Clearly these trials are subject to bias due to non-randomized selection, possible lack of generalizability to Canadian patients, and heterogeneous patient populations. Therefore, there is an important clinical need to investigate combined RT+TACE to improve outcomes in this rapidly growing poor prognosis patient population that has few options.

Research Design and Methodology The objective is to demonstrate superiority of SBRT in addition to TACE in terms of intrahepatic disease progression versus TACE alone using a randomized Phase III design. Phase I/II data has been published with recent data providing accurate event rates for statistical estimation of a small sample size requirement for this endpoint.

ELIGIBILITY:
Inclusion Criteria:

* HCC (diagnosed through biopsy or radiological criteria)
* Age >18 years of age
* Number of lesions: not more than 3 lesions
* Lesion size: up to 10 cm (and up to 10 cm cumulative diameter)
* Unilobar +/- segment 4
* Child-Pugh A within 6 weeks prior to study entry
* Barcelona Clinic (BCLC) Stage A/B
* Absence of comorbidities
* ECOG Performance Status 0-2
* Must be fit (eligible) for RT and TACE
* Unsuitable/unwilling for resection or transplant or radiofrequency ablation (RFA) or if these options are not available
* All blood work obtained within 6 weeks prior to study entry with adequate organ marrow function defined as follows:

Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 Platelets ≥ 50,000 cells/mm3 Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.) Total bilirubin < 2 mg/dL Prothrombin time/INR < 1.7 (unless on Coumadin/Warfarin) Albumin ≥ 28 g/L AST and ALT < 5 times ULN Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60 mL/min

* May have had previous surgery, ethanol injection and RFA to the liver
* No evidence of metastatic disease including nodal or distant metastases (clinically defined by each institution).
* Distance between GTV (lesion) and luminal structures (including esophagus, stomach, duodenum, small or large bowel) is >5 mm

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (Note that carcinoma in situ of the breast, oral cavity, or cervix are all permissible). No active cancer therapy.
* Major vascular invasion/thrombus
* Unsuitable for or refractory to transarterial hepatic chemo-embolization (TACE) Raoul et al (2011)
* Previous TACE and radiation to the liver (including SIRT )
* Life-threatening condition including untreated HIV and active hepatitis B/C
* Pregnancy or women of childbearing potential require a negative pregnancy test within 28 days

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic progression | 2 years
  Lesion growth as characterized by RECIST criteria

SECONDARY OUTCOMES:
Response rate - Modified RECIST criteria | 2 years
  Response of treated lesions using modified RECIST criteria
Local failure - within 1 cm from the original tumor volume | 2 years
  evidence of disease within 1cm of the tumor
Overall survival | 2 years
  overall survival percentage
Toxicity | 2 years
  Measured by NCI - CTC V4.0 at year 2
QoL-quality of life | 2 years
  EORTC QLQC30 at year 2

OTHER OUTCOMES:
Cost-benefit | 2 years
  costs of performing both treatments versus TACE alone
Extrahepatic failure | 2 years
  enumeration of number of cancers outside the liver

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lock, MD, Principal Investigator — University of Western Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Will be centrally registered data, freely shareable under contract as per ICMJE
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: available January 2018
Access Criteria: No access limitations

REFERENCES:
- [Background] Jacob R, Turley F, Redden DT, Saddekni S, Aal AK, Keene K, Yang E, Zarzour J, Bolus D, Smith JK, Gray S, White J, Eckhoff DE, DuBay DA. Adjuvant stereotactic body radiotherapy following transarterial chemoembolization in patients with non-resectable hepatocellular carcinoma tumours of >/= 3 cm. HPB (Oxford). 2015 Feb;17(2):140-9. doi: 10.1111/hpb.12331. Epub 2014 Sep 4. PMID 25186290